CLINICAL TRIAL: NCT00108394
Title: Osteopenia and Renal Osteodystrophy: Evaluation and Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-017-02S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2008-03

CONDITIONS: Osteopenia; Renal Osteodystrophy
Keywords: Uremia; Dialysis; Clinical Trials; Bone Diseases, Metabolic; adynamic bone disease; low bone turnover
MeSH Terms: conditions — Bone Diseases, Metabolic; Chronic Kidney Disease-Mineral and Bone Disorder; Uremia | interventions — Pamidronate

INTERVENTIONS:
Drug: pamidronate

SUMMARY:
The purpose of this study is to demonstrate whether pamidronate will preserve or increase bone mass in patients with adynamic bone disease, caused by low bone turnover.

DETAILED DESCRIPTION:
Detailed Summary: Bone disease has been a well-recognized complication of renal disease for over 100 years. Until the advent of dialysis, however, it was only another of the many dreadful complications of a fatal disease. Almost since the onset of dialysis, however, bone disease and calcium metabolism presented major difficulties to patients and physicians. Recently we reported that dialysis patients had an 8-fold increase in hip fracture rate, compared to the normal population. In younger dialysis patients (age 30-50 years) this risk was increased to nearly 100 fold. We have also noted a similar or even higher incidence of fracture in the transplant population. Low bone mass has been found in dialysis patients by ourselves and other investigators, a finding in the general population which predisposes to fracture. In the dialysis population, bone histologic studies done by us and others have reported the adynamic (low turnover) lesion in more than half of the dialysis population. This lesion is similar to what is seen in osteoporosis. Thus, dialysis patients, like osteoporotics, have low bone mass, low bone turnover, and a high fracture rate. In the osteoporotic patients, various bisphosphonates have been shown to inhibit bone resorption, increase bone mass and decrease fracture rate. The only bisphosphonate approved for use in patients with renal failure is pamidronate. This agent has not been used extensively in the general population because it must be given intravenously. This, together with the fact that pamidronate has a bone half-life of over 300 days, actually makes this drug a strong candidate for the treatment of patients with renal failure. In this investigation we propose using pamidronate in patients with renal failure to prevent bone loss and fracture. We will monitor bone mass by DEXA in patients to assess treatment response, assess bone histology in selected subjects, and collect data on fractures in the population.

Comparison: Subjects with normal or low parathyroid hormone (PTH) who receive dosing with pamidronate will be compared to similar subjects who receive placebo. Comparison groups will be randomly assigned and assignment will be blind.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis dependent for a minimum of 3 months
* Age greater than 18 years
* Low or normal bone turnover as defined by a mean intact PTH ≤400 pg/ml from a minimum of two values 6 months apart
* Informed consent

Exclusion Criteria:

* Mean serum aluminum levels > 20 mcg/L during 1 year prior to consent
* Documented dementia
* Comorbidity such that survival for >3 years is unlikely
* Use of steroids within 3 months of consent
* Use of bisphosphonates in previous 2 years
* Use of sex hormones (testosterone or estrogen) within 3 months of consent
* Mean calcium < 9.0 mg/dL during the two months prior to consent
* Peritoneal dialysis patients
* Body weight < 45 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2007-09

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States